CLINICAL TRIAL: NCT05011019
Title: Phase Ib Clinical Trial to Evaluate the Safety and Efficacy of AL2846 Capsules in Chinese Patients With Type I Neurofibromatosis (Neurofibromatosis and Malignant Peripheral Nerve Sheath Tumors)
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of AL2846 Capsules in Chinese Patients With Type I Neurofibromatosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: sponsor adjusts its research and development strategy
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL2846-Ib-01
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Neurofibromatosis and Malignant Peripheral Nerve Sheath Tumors
MeSH Terms: conditions — Neurofibromatoses; Neurofibrosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL2846 Capsules (Experimental): During the dose escalation phase, patients enrolled in the group will first receive a single fasting administration（AL2846 capsules 120-150mg，oral）. The observation period is 3 days. If dose-limited toxity (DLT) does not occur, they will continue to receive multiple consecutive fasting administrations (120mg-150mg，once a day，oral ),every 28 days as a treatment cycle.
  During the dose expansion phase, patients will receive multiple consecutive fasting administrations (AL2846 capsules，120mg-150mg, oral ), every 28 days as a treatment cycle.
  Interventions: Drug: AL2846 capsules

INTERVENTIONS:
Drug: AL2846 capsules — AL2846 is a multi-target receptor tyrosine kinase inhibitor.

SUMMARY:
AL2846 is a multi-target receptor tyrosine kinase inhibitor. The purpose of this study is to evaluate the safety and efficacy of AL2846 capsules in Chinese patients with type I neurofibromatosis (NF1) (neurofibromas and malignant peripheral nerve sheath tumors).

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily join the study and sign the informed consent form;
* Aged 18 to 75 years (when signing informed consent); Eastern cooperative oncology group（ ECOG） score: ≤2 ; patients with malignant peripheral nerve sheath tumors （MPNST）who are expected to survive ≥12 weeks;
* NF1 patients (including patients with MPNST) who are judged by the investigator as incomplete surgical resection, require systemic treatment, and have measurable lesions;

Note: NF1 diagnostic criteria meets at least one of the following:

1. Genetic examination confirmation: test positive for NF1 germline mutation in a Clinical Laboratory Improvement Amendments （CLIA）-certified laboratory (positive NF1 germline mutation must be confirmed by the central laboratory of this project, or an NF1 mutation test report issued by a CLIA-certified laboratory;
2. Clinical and imaging examination confirmation: According to the clinical National Institute of Health (NIH) consensus criteria, at least two of the following NF1 diagnostic criteria are met:

   1. Six or more café-au-lait macules (≥0.5cm in prepubertal patients or ≥1.5 cm in post pubertal patients)
   2. Freckling in axilla or groin
   3. ≥2 neurofibromas of any type, or ≥1 plexiform neurofibromas
   4. Optic glioma
   5. Two or more Lisch nodules
   6. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   7. A first-degree relative with NF1

      - Patients who are confirmed by direct measurement or according to the Response Evaluation Criteria in Solid Tumors（RECIST） 1.1 standard that there is at least one evaluable lesion, and the diameter of the lesion is greater than 3 cm, and the lesion can be seen in three consecutive sections;
      * The main organs function well and meet the following standards:

<!-- -->

1. Blood routine examination standard (no blood transfusion and no hematopoietic stimulating factor drugs used for correction within 7 days before the examination):

   a. White blood cell count (WBC) ≥3.5×109/L b. Hemoglobin (HGB) ≥90 g/L; c. The absolute value of neutrophils (NEUT) ≥ 1.5×109/L; d. Platelet count (PLT) ≥ 100×109/L.
2. The biochemical inspection shall meet the following standards:

   a. Albumin (ALB) ≥35g/L; b. Total bilirubin (TBIL) ≤ 1.5× the upper limit of normal (ULN), and patients with Gilbert syndrome are ≤ 2.5× ULN; c. Alanine-based transferase (ALT) and aspartate-based transferase (AST) ≤2.5×ULN; d. Serum creatinine (CR) ≤1.5×ULN or creatinine clearance (CCR) ≥50ml/min (application of standard Cockcroft-Gault formula);
3. The coagulation function test shall meet the following standards:

   International normalized ratio (INR)≤1.5×ULN (have not received anticoagulant therapy);
4. Thyroid function examination must meet the following standards:

Thyroid-stimulating hormone (TSH)≤ULN; if abnormal, Triiodothyronine （T3） and thyroxine（T4）levels should be examined, and T3 and T4 levels are normal.

5. Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.

- Female patients of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum pregnancy test within 7 days before study entry Negative, and must be a non-lactating subject; male patients should agree to adopt avoidance measures during the study period and within 6 months after the end of the study period;

- Patients enrolled in the second stage need to be pathologically confirmed to be enrolled in cohort 1, cohort 2 or cohort 3.

Exclusion Criteria:

* Combined diseases and medical history:

  1. Patients who have other malignant tumors within 3 years before the first medication or are currently suffering from other malignancies. The following two situations can be enrolled: other malignant tumors treated by a single operation; achieving 5 consecutive years of disease-free survival (DFS);

  2. With factors that affect oral medications (such as dysphagia, chronic diarrhea and intestinal obstruction, etc.)

  3. Unreliable toxic reactions higher than Common Terminology Criteria for Adverse Events(CTCAE) v5.0 level 1 caused by any previous treatment, excluding hair loss;

  4. Received major surgical treatment or obvious traumatic injury within 28 days before the first medication;

  5. Long-term unhealed wounds or fractures caused by surgery or trauma;

  6. Arterial/venous thrombosis occurred within 6 months before the first medication, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;

  7. With a history of psychotropic drug abuse and cannot be quit or have mental disorders;

  8. There are risk factors for prolonging the corrected QT interval（QTc）interval, such as uncorrectable hypokalemia, hereditary long QT syndrome, or taking drugs that prolong the QTc interval (mainly class Ia, Ic, and III antiarrhythmic drugs) ；

  9. Past or current retinal vein stenosis, retinal detachment, central retinal vein occlusion, glaucoma, grade 1 cataract, related symptoms caused by the disease are not considered as exclusion criteria;

  10. Interstitial pneumonia, including clinically significant radiation pneumonia;

  11. Patients with any severe and/or uncontrollable disease, including:
  1. Unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
  2. Suffering from grade ≥2 myocardial ischemia or myocardial infarction, arrhythmia (including male QTc ≥450 ms (male), QTc ≥470 ms (female)) and grade ≥2 congestive heart failure (New York Heart Association ( NYHA) classification, appendix 2);
  3. Active or uncontrolled serious infection (≥CTCAE v5.0 Grade 2 infection);
  4. Active hepatitis: hepatitis B reference: HBsAg is positive, and the HBV DNA test value exceeds the upper limit of normal; hepatitis C reference: HCV antibody is positive, and the HCV virus titer test value exceeds the upper limit of normal; Note: Those who meet the criteria for entry, hepatitis B surface antigen-positive or core antibody-positive patients, and hepatitis C patients need to continue antiviral therapy to prevent virus activation;
  5. Renal failure requiring hemodialysis or peritoneal dialysis;
  6. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  7. Poor diabetes control (fasting blood glucose (FBG)> 10 mmol/L);
  8. Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein quantification is confirmed to be >1.0 g;
  9. Those who suffer from epilepsy and need treatment;
* Tumor-related symptoms and treatment:

  1. Have received surgery, chemotherapy, radiotherapy or other anti-cancer therapies within 4 weeks before the first medication (the washout period will be calculated from the end of the last treatment); Note: Those who have received local radiotherapy in the past can be included in the group if the following conditions are met: the end of radiotherapy is more than 4 weeks from the beginning of the study treatment (brain radiotherapy is more than 2 weeks); and the target lesion selected for this study is not in the radiotherapy area; Or the target lesion is located in the radiotherapy area, but the progress has been confirmed.

  2. Have received National Medical Products Administration(NMPA) approved Chinese patent medicines with anti-tumor indications (including compound cantharidin capsules, Kangai injections, Kanglaite capsules/injections, Aidi injections, Brucea javanica oil injections). /Capsules, Xiaoaiping Tablets/Injections, Huachansu Capsules, etc.) treatment;
* Research and treatment related:

  1. Patients who have previously received one of the following treatments:

     a. Patients who have received NF1 drug treatment within 3 months before enrollment, and the related side effects have not yet recovered to below grade 1 (except for hair loss). Note: Patients who are receiving NF1 drug treatment must recover from the acute toxicity of the current NF1 treatment to less than or equal to Grade 1 (refer to CTCAE v5.0) before entering this study; b. Patients Received tipifarnib, pirfenidone, peg-interferon, sorafenib or other VEGFR inhibitor or biological treatments within 14 days before receiving study drug treatment ; c. Receiving strong Cytochrome P450 3A4 enzyme（CYP3A4） inhibitors (amprenavir, atazanavir, boceprevir, clarithromycin, cornivatan, delavirdine, diltiazem, erythromycin) within 14 days before receiving study drug treatment , Fursanavir, Indinavir, Itraconazole, Ketoconazole, Lopinavir, Mibefradil, Miconazole, Nefazodone, Nefinavir, Posaconazole, Ritonavir, saquinavir, tilarrevir, telithromycin, verapamil, voriconazole, etc.) or strong inducers (carbamazepine, felbamate, nevirapine, phenobarbital, phenytoin, Patients with primidone, rifabutin, rifampicin, rifapentin, etc.), except for external use on the skin;
  2. Unable to perform Magnetic Resonance Imaging(MRI) examination and/or there are contraindications for MRI examination, such as prosthesis, orthotics or orthodontics, which will interfere with the volume analysis of the target Plexiform neurofibroma( PN) on MRI;
* Patients who need to take more than the recommended dose of vitamin E daily;
* Patients who have participated within 4 weeks before the first medication and used other anti-tumor clinical trial drugs or wihtin 5 half-lives;
* According to the judgment of the investigator, there are situations that seriously endanger the safety of the patients or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Adverse event rate | :Baseline up to 96 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs)
objective response rate (ORR) | Baseline up to 96weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Phase II clinical recommended dose （RP2D） | Baseline up to 96 weeks
  recommended dose of Phase II clinical trial
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
PFS rate of one year | up to 96 weeks
  Rate of patients with PFS reaching one year among all patients
Overall Survival（OS） | assessed up to100 months
  From date of first administration of test drug until the date of death from any cause
Pain Scale (self-report form) | up to 96 weeks
  Self-report of pain in target tumor and other parts of body
Quality of life related scale（European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire version 3.0, EORTC QLQ-C30(V3)） | up to 96 weeks
  Questionnaires about the quality of life (including mental state, appetite state, sleep, etc.)
The patient's overall impression of the severity of symptoms (self-report) | up to 96 weeks
  Self-report on the severity of tumor pain, overall pain status, and tumor-related problems other than pain (vision, hearing, mobility, hearing, appearance, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, School of Medicine, Shanghai JiaoTong University, Shanghai, Shanghai Municipality, China